CLINICAL TRIAL: NCT06498960
Title: Pivotal Study to Evaluate the Safety and Effectiveness of the CereVasc® eShunt® System in the Treatment of Normal Pressure Hydrocephalus
Brief Title: Evaluation of the Safety and Effectiveness of the CereVasc® eShunt® System in Normal Pressure Hydrocephalus
Acronym: STRIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CereVasc Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN 0036
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Normal Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- eShunt System (Experimental): Endovascular placement of the eShunt Implant
  Interventions: Device: CereVasc eShunt System
- VP Shunt (Active Comparator): Surgical ventriculo-peritoneal shunt procedure
  Interventions: Device: VP Shunt

INTERVENTIONS:
Device: CereVasc eShunt System — The eShunt System consists of the following components:
  * eShunt Implant
  * eShunt Delivery Catheter and Transfer Tool
  * eShunt Anchor
  Other Names: eShunt System; eShunt Implant
  Arms: eShunt System
Device: VP Shunt — Control arm - VP shunt
  Arms: VP Shunt

SUMMARY:
Prospective, multi-center, randomized, controlled trial of the eShunt System in the treatment of patients with normal pressure hydrocephalus.

DETAILED DESCRIPTION:
The STRIDE study is a prospective, multi-center, randomized, controlled trial of the eShunt System in the treatment of patients with normal pressure hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria:

1. Patients ≥60 years old on the day of study informed consent
2. Patient or legally authorized representative is able and willing to provide written informed consent
3. History or evidence of gait impairment with a duration ≥3 months
4. Clinical presentation consistent with NPH including two or more of the clinical triad (i.e., history of gait disturbance, progressive mental deterioration, and urinary urgency or incontinence), together with all of the following:

   1. Brain MRI signs of ventricular enlargement disproportionate to cerebral atrophy (Evans' Index >0.3) and the absence of severe hippocampal atrophy,
   2. Pre-procedure spinal tap test or lumbar drain with subsequent gait disturbance improvement (Timed Up and Go Test) of at least 20%,
   3. CSF opening pressure ≥8 cmH2O,
   4. Baseline cognitive evaluation assessed by Montreal Cognitive Assessment (MoCA) test score ≥12
5. Patient is willing and able to attend all scheduled visits and comply with study procedures.
6. Confirmation of anatomy suitable for the eShunt procedure, as determined by evaluation of pre-procedure imaging (CT and MRI) and approved by an independent anatomical screening committee.

Exclusion Criteria:

Each subject may not:

1. Be unable to walk 10 meters (33 feet) with or without an assistive device
2. Be diagnosed with obstructive hydrocephalus
3. Have an active systemic infection or infection detected in CSF
4. Have had prior or existing shunts, endoscopic third ventriculostomy, or any previous surgical intervention for hydrocephalus
5. Demonstrate hypersensitivity or contraindication to heparin or radiographic contrast agents against which the subject cannot be adequately pre-medicated, desensitized or where no alternative is available
6. Have occlusion or stenosis of the internal jugular vein which would prohibit access to the IPS
7. Present with venous distension in the neck on physical exam
8. Have medical conditions associated with prolonged elevation of jugular venous pressure, including jugular vein stenosis or stricture, right sided heart failure, cirrhosis of the liver, arteriovenous fistulas in the arm for dialysis purposes, or an arterial venous fistula or malformation in the neck or brain
9. Have history of bleeding diatheses, coagulopathy or refuse to consent for blood transfusion in cases of emergency
10. Have had an ischemic stroke or transient ischemic attack within 180 days of eShunt procedure
11. Have documented evidence of a deep vein thrombosis superior to the popliteal vein
12. Have intrinsic blood clotting disorder
13. Have medical conditions requiring anticoagulation which is unable to be managed to allow for surgical procedure
14. Have presence of a posterior fossa tumor or mass
15. Have a life expectancy <1 year
16. Be currently participating in another interventional (drug, device, etc.) research project that may confound the results of this study.
17. Have established diagnosis of neurodegenerative diseases such as Parkinson's disease, Alzheimer's disease, or Lewy body dementia
18. Be diagnosed with schizophrenia or any psychiatric diagnosis (including depression) that may complicate outcome evaluation
19. Need an intracranial neurosurgical procedure within 180 days of study index procedure
20. Be unwilling or unable to comply with follow-up requirements
21. Have mRS of 0, 5, or 6

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 6 months
  The Primary Effectiveness Endpoint of this study is change in gait impairment at 6-months, compared to baseline. Change in gait impairment is defined as reduction in time required to complete the Timed Up and Go (TUG) test (stand up, walk 3m, turnaround, walk 3m, sit down).
Primary Safety Endpoint | 6 months
  All adverse events will be reported for the investigational (eShunt System) and control (VP shunt) arms. Safety will be analyzed based on a review of all AEs in the investigational arm compared to the control arm, through 6-months post-procedure to demonstrate an acceptable safety profile of the eShunt System.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (26):
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Baptist Medical Center - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health, West Bloomfield, Michigan
  - Cooper Neurological Institute, Camden, New Jersey
  - Albany Medical Center, Albany, New York
  - University at Buffalo Neurosurgery, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Virginia Commonwealth University, Richmond, Virginia
- Clinica La Sagrada Familia, Buenos Aires, Argentina
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No